CLINICAL TRIAL: NCT00790751
Title: A Randomized, Double-Blind, Placebo-Controlled Evaluation of the Safety and Efficacy of Avanafil (TA-1790) in Subjects With Generalized Erectile Dysfunction
Brief Title: Research Evaluating an Investigational Medication for Erectile Dysfunction - General ED
Acronym: REVIVE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: VIVUS LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TA-301
Record Dates: First submitted 2008-11-10; First posted 2008-11-13 (Estimated); Results first posted 2012-06-28 (Estimated); Last update posted 2012-07-11 (Estimated); Status verified 2012-06

CONDITIONS: Erectile Dysfunction
Keywords: ED; Erectile Dysfunction; Dysfunction; Erectile
MeSH Terms: conditions — Erectile Dysfunction | interventions — avanafil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- placebo (Placebo Comparator)
  Interventions: Drug: placebo
- avanafil 50 mg (Experimental)
  Interventions: Drug: avanafil
- avanafil 100 mg (Experimental)
  Interventions: Drug: avanafil
- avanafil 200 mg (Experimental)
  Interventions: Drug: avanafil

INTERVENTIONS:
Drug: placebo — 30 minutes orally prior to initiation of sexual activity
  Arms: placebo
Drug: avanafil — 30 minutes orally prior to initiation of sexual activity
  Other Names: TA-1790; Stendra
  Arms: avanafil 50 mg
Drug: avanafil — 30 minutes orally prior to initiation of sexual activity
  Other Names: TA-1790; Stendra
  Arms: avanafil 100 mg
Drug: avanafil — 30 minutes orally prior to initiation of sexual activity
  Other Names: TA-1790; Stendra
  Arms: avanafil 200 mg

SUMMARY:
This study is being conducted to compare the safety and efficacy of 3 doses of avanafil to placebo in men with mild to severe erectile dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* Male subjects, age ≥ 18 years;
* Minimum 6 month history of mild to severe erectile dysfunction;
* Subject is in a monogamous, heterosexual relationship for at least 3 months;
* Subject agrees to make at least 4 attempts at intercourse per month;
* Subject is willing and able to provide informed consent.

Exclusion Criteria:

* Allergy or hypersensitivity to PDE5 inhibitors;
* History of dose-limiting AEs during therapy with a PDE5 inhibitor or hx of consistent treatment failure with other PDE5 inhibitors for therapy of ED;
* Current or expected use of organic nitrates at any time during the study;
* Previous or current antiandrogen therapy;
* Use of prescription or over-the-counter drugs known to inhibit the activity of CYP3A4 at any time during the study;
* Androgen replacement therapy that has not been stable for at least 3 month;
* Initiation or change in dose of any alpha-blocker within 14 days prior to randomization;
* ED as a result of spinal cord injury or radical prostatectomy;
* Untreated hypogonadism or low serum total testosterone
* History of or predisposition to priapism;
* Any penile implant;
* Elevated PSA, other evidence of prostate cancer, or previous radical prostatectomy;
* History of any malignancy (except basal cell carcinoma or squamous cell carcinoma of the skin successfully treated by curative excision);
* History of type 1 or type 2 diabetes;
* Uncontrolled hypertension;
* Hypotension;
* Orthostatic hypotension;
* Significant cardiovascular disease;
* Abnormal ECG;
* Hepatic or renal impairment;
* Positive STD screen;
* Clinically evident penile lesions, abrasions, or anatomical deformities;
* Urinary tract or bladder infection;
* Use of any treatment for erectile dysfunction other than study drug at any time during the study;
* Participation in another investigational study within 30 days of screening or at any time during this study;
* Previous participation in any other investigational study of avanafil;
* History or current drug, alcohol, or substance abuse;
* Any history of bipolar disorder or psychosis, greater than one lifetime episode of major depression, current depression of moderate or greater severity or antidepressant use that has not been stable for at least 3 months;
* Partners who are < 18 years of age, who are nursing, who are known to be pregnant at screening, who wish to become pregnant during the study period, who have any gynecologic problems or major medical conditions that would limit participation in sexual intercourse;
* Evidence of any other condition by history, physical examination, or laboratory studies that, in the opinion of the investigator, would contraindicate the administration of study medication, affect compliance, interfere with study evaluations, limit study participation, contraindicate sexual activity, or confound the interpretation of study results.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 646 (Actual)
Dates: Start 2008-11; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Irwin Goldstein, MD, Principal Investigator — San Diego Sexual Medicine
Locations (36):
- United States (36):
  - Research Site, Birmingham, Alabama
  - Research Site, Homewood, Alabama
  - Research Site, Tucson, Arizona
  - Research Site, Sacramento, California
  - Research Site, San Diego, California
  - Research Site, Waterbury, Connecticut
  - Research Site, Clearwater, Florida
  - Research Site, Coral Gables, Florida
  - Research Site, Hialeah, Florida
  - Research Site, Jacksonville, Florida
  - Research Site, Jupiter, Florida
  - Research Site, Ocala, Florida
  - Research Site, Pembroke Pines, Florida
  - Research Site, Tampa, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Wichita, Kansas
  - Research Site, Madisonville, Kentucky
  - Research Site, Shreveport, Louisiana
  - Research Site, Kansas City, Missouri
  - Research Site, Lawrenceville, New Jersey
  - Research Site, Albany, New York
  - Research Site, New York, New York
  - Research Site, Cary, North Carolina
  - Research Site, Charlotte, North Carolina
  - Research Site, Harrisburg, North Carolina
  - Research Site, Hickory, North Carolina
  - Research Site, Raleigh, North Carolina
  - Research Site, Salisbury, North Carolina
  - Research Site, Wilmington, North Carolina
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Beachwood, Ohio
  - Research Site, Bala-Cynwyd, Pennsylvania
  - Research Site, Lancaster, Pennsylvania
  - Research Site, El Paso, Texas
  - Research Site, Houston, Texas
  - Research Site, Spring, Texas

REFERENCES:
- [Result] Goldstein I, McCullough AR, Jones LA, Hellstrom WJ, Bowden CH, Didonato K, Trask B, Day WW. A randomized, double-blind, placebo-controlled evaluation of the safety and efficacy of avanafil in subjects with erectile dysfunction. J Sex Med. 2012 Apr;9(4):1122-33. doi: 10.1111/j.1743-6109.2011.02629.x. Epub 2012 Jan 16. PMID 22248153

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subject recruitment occurred at US investigative sites between November 2008 and April 2009.
Pre-assignment Details: Subjects meeting the initial eligibility criteria completed a 4-week non-treatment run-in period during which information on each attempt at intercourse was recorded. At the end of the run-in, subjects meeting the randomization criteria were eligible for assignment to one of the treatment groups.
Groups:
- Placebo: placebo 30 minutes orally prior to initiation of sexual activity
- Avanafil 50 mg: avanafil 50 mg 30 minutes orally prior to initiation of sexual activity
- Avanafil 100 mg: avanafil 100 mg 30 minutes orally prior to initiation of sexual activity
- Avanafil 200 mg: avanafil 200 mg 30 minutes orally prior to initiation of sexual activity
Period: Overall Study
Arm/Group | Placebo | Avanafil 50 mg | Avanafil 100 mg | Avanafil 200 mg
Started | 162 | 161 | 161 | 162
Completed | 137 | 131 | 141 | 141
Not Completed | 25 | 30 | 20 | 21
Not completed — Protocol non-compliance | 16 | 16 | 10 | 11
Not completed — Lost to Follow-up | 4 | 9 | 4 | 5
Not completed — Adverse Event | 5 | 3 | 5 | 4
Not completed — Requirement for restricted medication | 0 | 2 | 0 | 0
Not completed — Death | 0 | 0 | 1 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Avanafil 50 mg | Avanafil 100 mg | Avanafil 200 mg | Total
Number analyzed (Participants) | 162 | 161 | 161 | 162 | 646
Age Continuous [Mean (Standard Deviation); unit: years] | 55.4 (11.13) | 55.4 (10.81) | 56.5 (10.32) | 55.7 (11.33) | 55.7 (10.89)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0
  Male | 162 | 161 | 161 | 162 | 646
Region of Enrollment [Number; unit: participants]
  United States | 162 | 161 | 161 | 162 | 646

OUTCOME MEASURES:

1. Primary Outcome: Change in Percentage of Sexual Attempts in Which Subjects Were Able to Maintain an Erection of Sufficient Duration to Have Successful Intercourse
Description: Data presented as mean change from baseline in the percentage of Yes responses to Sexual Encounter Profile (SEP) diary question 3 "Did your erection last long enough for you to have successful intercourse?"
Time Frame: Baseline, 12 weeks
Population: Number of participants analyzed represents the Intent-to-Treat population.
Measure: Least Squares Mean (Standard Error); unit: percentage of sexual attempts
Arm/Group | Placebo | Avanafil 50 mg | Avanafil 100 mg | Avanafil 200 mg
Number analyzed (Participants) | 155 | 154 | 157 | 156
percentage of sexual attempts | 14.1 (2.57) | 27.8 (2.58) | 43.4 (2.56) | 44.2 (2.57)

2. Primary Outcome: Change in Percentage of Sexual Attempts in Which Subjects Were Able to Insert the Penis Into the Partner's Vagina
Description: Data presented as mean change from baseline in the percentage of Yes responses to Sexual Encounter Profile (SEP) diary question 2 "Were you able to insert your penis into your partner's vagina?"
Time Frame: Baseline, 12 weeks
Population: Number of participants analyzed represents the Intent-to-Treat population.
Measure: Least Squares Mean (Standard Error); unit: percentage of sexual attempts
Arm/Group | Placebo | Avanafil 50 mg | Avanafil 100 mg | Avanafil 200 mg
Number analyzed (Participants) | 155 | 154 | 157 | 156
percentage of sexual attempts | 7.1 (2.33) | 18.2 (2.34) | 27.2 (2.32) | 29.8 (2.33)

3. Primary Outcome: Change in International Index of Erectile Function - Erectile Function Domain (IIEF-EF) Score
Description: Questionnaire assesses subject's evaluation of erectile function over the previous 4-week period. Total score from questions 1-5 & 15 ranges from 1 to 30. A higher score indicates better erectile function.
Time Frame: Baseline, End of Treatment (up to 12 weeks)
Population: Number of participants analyzed represents the Intent-to-Treat population. For dropouts or missing data, the last observation carried forward convention was used.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | Avanafil 50 mg | Avanafil 100 mg | Avanafil 200 mg
Number analyzed (Participants) | 152 | 152 | 156 | 155
scores on a scale | 2.9 (0.57) | 5.4 (0.57) | 8.3 (0.56) | 9.5 (0.56)

ADVERSE EVENTS:
Time Frame: AE reporting began when the subject provided written informed consent and extended until 28 calendar days after the last dose of the investigational product was administered, or until the subject was discontinued from the study, whichever was later.
Description: # participants at risk is presented for the safety population. The Safety Population was defined as all subjects who took at least one dose of study drug and had safety data available.
Arm/Group | Placebo | Avanafil 50 mg | Avanafil 100 mg | Avanafil 200 mg
Serious Adverse Events (participants affected / at risk) | 2/161 | 1/160 | 3/161 | 3/162
Other Adverse Events (participants affected / at risk) | 7/161 | 16/160 | 28/161 | 31/162
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=161) | Avanafil 50 mg (N=160) | Avanafil 100 mg (N=161) | Avanafil 200 mg (N=162)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Prostate cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infected bites (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gun shot wound (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Depression suicidal (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=161) | Avanafil 50 mg (N=160) | Avanafil 100 mg (N=161) | Avanafil 200 mg (N=162)
Nasopharyngitis (Infections and infestations) | 2 | 1 | 2 | 6
Bronchitis (Infections and infestations) | 1 | 3 | 1 | 4
Headache (Nervous system disorders) | 2 | 7 | 12 | 15
Flushing (Vascular disorders) | 0 | 6 | 10 | 6
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 7 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After Sponsor's written notification that publication of results is no longer planned or 12 months after termination of the study at all sites, Institution & PI may publish, upon written approval from Sponsor, results of the Study. Sponsor will be given the opportunity to review any proposed publication at least 60 days prior to submission for publication or disclosure. Upon Sponsor's written request, Institution and PI shall not publish or disclose information related to the Study.